CLINICAL TRIAL: NCT01537731
Title: Chronic Pain After Vaginal or Laparoscopic Hysterectomy for Benign Conditions
Brief Title: Vaginal or Laparoscopic Hysterectomy, Persistent Postsurgical Pain
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Arvi Yli-Hankala, professor, Tampere University Hospital
Other Study IDs: R08031M R09003
Record Dates: First submitted 2012-01-10; First posted 2012-02-23 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hysterectomy: Patient who previously underwent vaginal or laparoscopic hysterectomy
  Interventions: Procedure: vaginal or laparoscopic hysterectomy

INTERVENTIONS:
Procedure: vaginal or laparoscopic hysterectomy — vaginal hysterectomy or laparoscopic hysterectomy

SUMMARY:
Previous studies have shown that chronic pain after hysterectomy is common. The aim of this study is to investigate the incidence of chronic pain after vaginal or laparoscopic hysterectomy for benign reasons. The aim of this prospective study is also to study the role of anesthetics, surgery and other possible predictors for pain 6 months after hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo vaginal or laparoscopic hysterectomy for benign conditions
* Age 18-69 years
* Gender: female
* ASA status 1-3

Exclusion Criteria:

* Body Mass Index over 35
* Diabetes mellitus
* Liver disease
* Preoperative use of opioids

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who undergo vaginal or laparoscopic hysterectomy for benign conditions.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Presence of persistent postsurgical pain as measured at 6 months after surgery. | five years

SECONDARY OUTCOMES:
Severity, location, characteristics of persistent postsurgical pain. | five years
Effect of postsurgical pain on activity, sleep. | five years

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Pokkinen SM, Nieminen K, Yli-Hankala A, Kalliomaki ML. Persistent posthysterectomy pain: A prospective, observational study. Eur J Anaesthesiol. 2015 Oct;32(10):718-24. doi: 10.1097/EJA.0000000000000318. PMID 26258656